CLINICAL TRIAL: NCT04942782
Title: Lumbopelvic Stabilization Versus Pilates Exercises On Gait Cycle Phases And Maximum Peak Pressure On Foot In Chronic Nonspecific Low Back Pain: Randomized Controlled Trial
Brief Title: Lumbopelvic Stabilization Versus Pilates Exercises On Gait Phases And Peak Pressure On Foot In Low Back Pain
Acronym: LBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p.t.REC/012/003225
Record Dates: First submitted 2021-06-24; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Low Back Pain
Keywords: lumbopelvaic stabilization exercise; pilates exercise; gait cycle phases; peak pressure
MeSH Terms: conditions — Low Back Pain | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: lumbopelvic stabilization and Pilates
Who Masked: Participant, Outcomes Assessor
Masking Description: random generator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lumbopelvic stabilization exercises (Experimental): the patients will receive trunk stabilization exercise +strengthening exercises for the abdominal, back, and hip muscles three times/ week for three months
  Interventions: Other: lumbopelvic stabilization exercises; Other: conventional therapy
- Pilates exercises (Experimental): the patients will receive trunk pilates exercise +strengthening exercises for the abdominal, back, and hip muscles three times/ week for three months
  Interventions: Other: pilates exercise; Other: conventional therapy
- conventional therapy (Active Comparator): the patients will receive trunk stabilization exercise three times/ week for three months
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: lumbopelvic stabilization exercises — the patients will receive lumbopelvic stabilization in the form of three parts: 1 Segmental control over primary stabilizers (mainly TrA, deep multifidus, pelvic floor and diaphragm) 2-Exercises in closed chain, with low velocity and low load 3-Exercises in open chain, with high velocity and load
  Arms: lumbopelvic stabilization exercises
Other: pilates exercise — the patient will receive pilates exercise in the form of Breast stroke prep, Side leg lift series, One leg circle, Hundreds, Shoulder bridge, and Spine stretch forward
  Arms: Pilates exercises
Other: conventional therapy — Patients will received strengthening exercises for the abdominal, back, and hip muscles. The patients performed an average of three series of ten repetitions of each exercise. Increases in the number of exercises performed in each session (or load progression) occurred according to individual tolerance

SUMMARY:
the purpose of this trial is to investigate and compare between lumbopelvic stabilization and pilates exercises on gait cycle phases and maximum peak pressure on the foot in chronic nonspecific low back pain?

DETAILED DESCRIPTION:
LBP is the leading cause of activity limitation, results in significant losses in productivity at work, and incurs billions of dollars in medical expenditure annually So, the aim of physical therapy treatment in the patient with chronic nonspecific low back pain is more effective in improving gait cycle phases and maximum peak pressure on the foot and help LBP patients to walk normally as much as possible, also this will improve our body of knowledge about the best modalities for treating LBP. The finding of this study may help LBP patients avoid exposure to complications due to altered gait cycle phases and maximum peak pressure on the foot. Also, it will help physiotherapists to know which treatment will be effective in improving gait cycle phases and maximum peak pressure on the foot. one hundred patients with mechanical low back pain will be allocated randomly to three groups; group A will receive pilates, group B will receive lumbopelvic stabilization exercise and group C will receive strengthening exercises for the abdominals, back, and hip muscles

ELIGIBILITY:
Inclusion Criteria:

1. Their age between 20 and 40 years
2. patients is required to have chronic nonspecific LBP (more than12 weeks), deﬁned as Pain in the lumbar and/or buttock region (defined as pain reported below the level of T12 and no lower than the buttock line).
3. Patients will be excluded if they have signs of serious spinal pathology (red flags) including significant trauma, unexplained weight loss, and widespread neurologic changes

Exclusion Criteria:

1. subjects with specific back pain (fracture, osteoporosis or degenerative changes, prolapse intervertebral disc, bone disorders, arthritis, tumour),
2. subjects with neurological involvement (radiculopathy, myelopathy),
3. subjects with previous spinal surgery

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
gait cycle phases and maximum peak pressure on foot | up to twelve weeks
  gait cycle phases and peak pressure will be measure by Tekscan walkway

SECONDARY OUTCOMES:
pain intensity | up to twelve weeks
  visual analogue scale will be used for measuring pain level
disability | up to twelve weeks
  Functional disability of each patient was assessed by Modified Oswestry Disability Questionnaire
muscle endurance | up to twelve weeks
  Sorensen test (low back fatigue test) and Trunk flexion endurance test will be used for measuring the level of endurance